CLINICAL TRIAL: NCT01814839
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single- and Multi-Dose, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered ALN-TTRSC in Healthy Volunteers
Brief Title: A Phase 1, Single- and Multi-Dose, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered ALN-TTRSC (Revusiran) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-TTRSC-001
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: TTR-mediated Amyloidosis
Keywords: RNAi therapeutic
MeSH Terms: interventions — revusiran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-TTRSC (revusiran) (Active Comparator)
  Interventions: Drug: ALN-TTRSC (revusiran)
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-TTRSC (revusiran) — Ascending doses of ALN-TTRSC (revusiran) by subcutaneous (SC) injection
  Arms: ALN-TTRSC (revusiran)
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of ALN-TTRSC (revusiran) in healthy volunteer subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) must be ≥ 16.5 kg/m2 and ≤ 35.0 kg/m2;
* Female subjects must be of non-childbearing potential; e.g., postmenopausal or pre-menopausal with surgical sterilization;
* Male subjects agree to use appropriate contraception;
* Adequate blood counts, liver and renal function;
* Non-smokers for at least 3 months;
* Willing to give written informed consent and are willing to comply with the study requirements;
* Subject was born in Japan and has lived outside of Japan for <10 years, and subject's biological parents and grandparents are fully Japanese and were born in Japan (cohorts 19 and 20).

Exclusion Criteria:

* Known human immunodeficiency virus (HIV) positive status or known or suspected systemic bacterial, viral, parasitic, or fungal infection;
* Subjects with a history of multiple drug allergies or intolerance to SC injection;
* History of drug abuse and/or alcohol abuse;
* Receiving an investigational agent within 3 months prior to study drug administration;
* Considered unfit for the study by the Principal Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs) and study drug discontinuation. | Up to 63 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ALN-TTRSC (revusiran) (Cmax, tmax, t1/2, AUC0-last, CL). | Up to 90 days
Effect of ALN-TTRSC (revusiran) on transthyretin (TTR) (Determination of % Lowering of TTR to pretreatment/Baseline Levels). | Up to 90 days
Effect of ALN-TTRSC (revusiran) on vitamin A (Determination of % Lowering of vitamin A to pretreatment/Baseline Levels). | Up to 90 days
Effect of ALN-TTRSC (revusiran) on retinol binding protein (RBP) (Determination of % Lowering of RBP to pretreatment/Baseline Levels). | Up to 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Clinical Site, Leeds
  - Clinical Site, London